CLINICAL TRIAL: NCT04080115
Title: A Randomized Controlled Trial Examining the Impact of a Brief Attention-based Neurobehavioral Transdiagnostic Intervention on Acute Fear Response
Brief Title: Does Increasing Attentional Control Decrease Acute Fear Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-382
Record Dates: First submitted 2019-08-21; First posted 2019-09-06 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Fear; Attention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Training Technique (ATT) (Experimental)
  Interventions: Behavioral: Attention Training Technique
- Sham intervention control condition (Active Comparator)
  Interventions: Behavioral: Sham intervention control condition

INTERVENTIONS:
Behavioral: Attention Training Technique — ATT will be administered through a customized Expiwell smartphone application that will be downloaded onto participants' cell phones at the first laboratory session (T2). For the purposes of the proposed study, participants need to complete the intervention once a day, for the six days between their lab sessions; signals will begin the day after their T2 session and they will be notified up to a maximum of five times per day to complete their daily session. The ATT sessions are comprised of three phases. The first is a 5-minute phase during which the participant is instructed to attend to specific sounds in the recording and disregard other sounds. The subsequent 5-minute phase includes instructions to rapidly switch their attention between sounds in the recording. The final phase is a dual attention task lasting 2 minutes wherein the participant is instructed to pay attention to multiple sounds in the recording at once. In total, each session of ATT lasts 12 minutes.
  Arms: Attention Training Technique (ATT)
Behavioral: Sham intervention control condition — The sham control condition consists of the same 12 minutes of simultaneous sounds as the ATT technique, but will not include any verbal instruction, thus isolating the effects of intentional orientation of attention.
  Arms: Sham intervention control condition

SUMMARY:
Despite decades of research, current psychological treatments designed to treat a variety of mental illnesses are not effective for all who receive them. Specifically, well-supported treatments for mental illnesses that involve fear (e.g., PTSD, panic) appear to be effective for the majority of individuals, but consistently leave a group of "treatment non-responders." One potential explanation for the observed discrepancy in treatment response may be the focus of modern psychotherapies on relieving symptoms specific to categorical diagnoses, rather than mechanisms underlying why the individual is experiencing the symptoms. Recently, fear-based psychological disorders (e.g., PTSD, specific phobia, panic disorder, social anxiety) have been identified as sharing a distinct set of biomarkers, including genetic biomarkers of acute fear (i.e., fear in the moment) and impairments in controlling attention. Neurobehavioral interventions are therefore a promising class of treatments designed to target the biological markers that may be maintaining the symptoms of various psychological disorders. The Attention Training Technique (ATT) is a neurobehavioral intervention that has garnered attention through its demonstrated effectiveness in reducing symptoms across a variety of psychological diagnoses. While grounded in well-established theory, the mechanisms of change in ATT are largely unknown. One proposed mechanism may be that ATT promotes functional connectivity between regions in the brain implicated in top-down executive control over attention (ventromedial prefrontal cortex [vmPFC] and dorsolateral prefrontal cortex [dlPFC]) and bottom-up attention networks (dorsal anterior cingulate cortex [dACC] and amygdala), resulting in increased top-down regulation of potentially problematic bottom-up attentional processes. The same brain regions implicated in both top-down and bottom-up attentional processes have also been associated with fear responding (i.e., startle response) and fear learning (i.e., how quickly one learns that a stimuli is safe or to be feared). Taken together, the research suggests that acute fear responding may be decreased through increased executive control over attention through engagement in ATT. The proposed randomized clinical trial will test whether a self-administered brief neurobehavioral intervention (ATT) to increase attentional control will decrease acute fear responding, and whether this change is associated with increased ability to handle attentional interference, an ability associated with normative dACC functioning and measured by behavioral proxy in this study via the Multi-Source Interference Task (MSIT). It is expected that those who engage in ATT will show greater attentional control efficiency, which will decrease their acute fear response. It is also expected that those who engage in ATT will also show lower sensitivity to attentional interference (measured through the MSIT) and will exhibit decreases in their reported fear as their attentional control increases over the course of the intervention. Additionally, it is expected that the intervention (ATT) will indirectly decrease symptoms of categorical fear-based psychological diagnoses through the identified biomarkers (i.e., attentional control, attentional interference sensitivity, acute fear response) to decrease reported symptoms.

DETAILED DESCRIPTION:
Participants will be directed to complete the T1 survey within the week before the first session of the multi-session study. The T1 survey will assess symptoms of fear-based psychological disorders, attentional control, autonomic arousal and threat perception. Additionally, participants will complete a flanker task.

At the first laboratory session, participants will complete the Attention Network Task (ANT), the Fear Potentiated Startle (FPS) paradigm and the Multi-Source Interference Task (MSIT). Participants will be prepared for the protocol through affixing two 5 mm Ag/AgCl pre-gelled disposable electrodes approximately 1 cm under the pupil and 1 cm below the lateral canthus to assess electromyography of the orbicularis oculi muscle contraction for the FPS paradigm, and all resistance will be kept less than 6 kΩ.

Following the resting phase, the FPS paradigm will begin. For the proposed study, the aversive unconditioned stimulus (US) will be a 250-ms airblast with an intensity of 140 p.s.i. directed to the larynx. The conditioned stimuli (CS) consist of different colored shapes presented on a computer monitor utilizing SuperLab 4.0 for Windows (Cedrus, Inc.). The startle probe will be comprised of a 108 A-weighted decibel 40-ms burst of broadband noise with near instantaneous rise, which is presented via headphones after 6 s and will be followed by the US 0.5 s later. The CS+ will be paired with the airblast, while the CS- will not. Fear-potentiation and extinction occur across two active phases. The first 20 minute phase includes fear acquisition. During this period, a colored shape will be the reinforced conditioned stimulus (CS+) through its association with the aversive US. A second shape, the non-reinforced conditioned stimulus (CS-), and noise probe alone (NA) will also be presented. The conditioning phase includes three blocks of four trials of each type of stimulus (i.e., NA, CS+, CS-) in each block. All trials in both phases are presented on a fixed schedule with inter-trial intervals ranging between 18 and 25 seconds. Upon conclusion of the acquisition phase, participants complete the MSIT before beginning the extinction phase.

Following the completion of the MSIT, a 25-minute extinction phase begins. The extinction phase will consist of five blocks of four trials of each type (NA, CS+ [unreinforced], and CS-) in each block. Throughout the FPS paradigm, participants are asked to use a keypad to press a button marked "+" if they expect a CS to be followed by the US, a button marked "-" if they do not expect a CS to be followed by the US, and a button marked "0" if they are uncertain of what to expect. Following the FPS paradigm at T2, participants will download and learn to use the study application, whereas at T4, participants will complete the computerized post-intervention survey (same as baseline survey).

Over the course of the next 6 days following T2, participants will complete 6 sessions of the ATT or the sham control condition when prompted by the Expiwell app on their smartphone. Upon completion of the intervention, participants will complete a short assessment of their self-reported attentional control and experience of fear since the last signal. Exactly one week from the first laboratory session (i.e., same day of the week, same time of day) participants will return to the laboratory for the second lab session (T4). Participants will complete informed consent, followed by ANT, FPS, and MSIT paradigms. Upon completion of the FPS paradigm, participants will complete a computerized survey that includes measures of fear-related symptomatology and attentional control that will be modified to assess experiences over the past week. One month following the final lab session (T4), participants will be emailed the follow-up survey (T5) The T5 survey assesses fear-related symptomatology over the past month since T4.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled student at Northern Illinois University
* Age at least 18 years old
* fluent in English
* Elevated symptoms of a fear-based disorder (i.e., PTSD, social anxiety, panic, specific phobia; Gorka et al., 2017)
* Increased reaction times on flanker task
* Possession of an Android or IOS smartphone

Exclusion Criteria:

* auditory or visual impairment
* active psychotic symptoms
* self-reported diagnosis of ADHD including a prescription for stimulant medication for the treatment of ADHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Attention Network Task(ANT)/Attentional Control Efficiency at Post-intervention | Day 1 (Baseline/pre-intervention) and Day 7 (Post-intervention)
  The ANT is a behavioral reaction time (RT) measure of attentional alerting, orienting, and executive control (Fan et al., 2002). The test is a combination of the commonly used flanker task (see Eriksen & Eriksen, 1974) and a simple cued reaction time task (see Posner, 1980). The ANT provides measures of both RT and error rates (ER). There are several test conditions of interest in the ANT that produce scores that are indications of efficiency in the three separate attention networks.
Change in Acute Fear Response (i.e., Fear Load and Fear Inhibition) at Post-intervention | Day 1 (Baseline/pre-intervention) and Day 7 (Post-intervention)
  The acoustic startle response (eyeblink component) will be measured via electromyography (EMG) of the right orbicularis oculi muscle and will be measured as the maximum amplitude of the eyeblink muscle contraction 20 to 200 ms after the startle probe is presented. FPS score will be calculated by subtracting startle magnitude to the noise alone trials (NA) from the startle magnitude to the CS in each conditioning block. For the purposes of the current study, acute fear is conceptualized as fear load and fear inhibition. Fear load will be operationalized as the FPS score to the CS+ during the first and second blocks of the extinction phase and fear inhibition is operationalized as the FPS to CS+ in the last two blocks of extinction. Fear load and fear inhibition are continuous scores when calculated in such a manner.
Change in dACC functioning, as measured by a behavioral proxy (i.e., Multi-Source Interference Task) | Day 1 (Baseline/pre-intervention) and Day 7 (Post-intervention)
  The Multi-Source Interference Task (MSIT; Bush, Shin, Holmes, Rosen & Vogt, 2003) is a behavioral task designed to cognitively tax the cingulo-frontal parietal cognitive/attention network with two conditions (i.e., interference and control) and two performance scores (i.e., absolute and relative processing speed). Specifically, in an fMRI study, Bush and colleagues (2003) showed that the MSIT activates the dACC, specifically, to a greater degree than any previously utilized behavioral task.
Change in Self-Reported Attentional Control:. Attentional Control Scale, Short form (ACS-S; Judah et al., 2014) | Day 0 (Online baseline survey) through study completion, anticipated average 6 weeks
  The ACS-S form is a 12-item short form of the Attentional Control Scale (Derrybery & Reed, 2002). Similar to the long form, the ACS-S measures perceived attentional control, consisting of attentional focusing (i.e., When I am reading or studying, I am easily distracted if there are people talking in the same room) and attention shifting (i.e., It is easy for me to alternate between two different tasks). Participants rate their agreement with each item on a 1 (Almost never) to 4 (Always) scale as each statement applies to them. Higher scores reflect greater perceived attentional regulation.
Change in Self-reported Fear: NIH Toolbox for Assessment of Neurological and Behavioral Function- Fear (NIHTB- Fear; Salsman et al., 2013) | Day 0 (Online baseline survey) through study completion, anticipated average 6 weeks
  The Fear-Affect survey is a 29-item measure of symptoms of anxiety that reflect the presence of autonomic arousal (e.g., I had a racing or pounding heart) and threat perception (e.g., I felt fearful). Participants rate their agreement with a 7-day timeframe for each item on a 5-point Likert scale from 1 (Never) to 5 (Always), with higher scores reflecting more fearful responding; a T score of 60 is recommended as the cut-off for high levels of fear responding (Slotkin et al., 2012), and as such will serve as the cut-off for inclusion criteria in the proposed study. The short form of the Fear Affect scale will also be utilized by the proposed study during the Ecological Momentary Assessment (EMA) intervention period (T3). The Fear-Affect short form is a 7-item measure assessing fearful emotions in the past 7 days on the same 5-point Likert scale. For T3, the time frame will be "since the last signal." For T5, the time frame will be modified to "in the past month."

SECONDARY OUTCOMES:
Change in Panic Disorder Self-Report (PDSR; Newman, Holmes, Zuellig, Kachin & Behar, 2006) | Day 0 (Online baseline survey), Day 7, and one month follow-up (week 5)
  The PDSR is a brief 24-item measure of panic disorder (PD) originally designed based on the Diagnostic and Statistical Manual, 4th edition (APA, 1994). The initial items assess if participants have experienced a panic attack as defined as a "sudden rush of intense fear or anxiety," and if so, recency and frequency of the attack(s). If lifetime panic attacks exceed 1 attack, presence of physiological symptoms, fear of dying and losing control, as well as functional impairment and distress related to the panic attacks are assessed. The PDSR has demonstrated strong psychometric properties, with good test-retest reliability high internal consistency, and discriminant and convergent validity in the original validation study (Newman et al., 2006). A diagnostic cut-off score of 8.75 has demonstrated high agreement with a diagnostic interview in identifying those who meet criteria for PD (k = .93; Newman et al., 2006). For T4, the time frame will be modified to "In the last 7 days."
Change in Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998) | Day 0 (Online baseline survey), Day 7, and one month follow-up (week 5)
  The SIAS is a 20-item self-report measure of anxiety in social interactions, both in dyadic (e.g., I feel tense if I am alone with just one other person) and group settings (e.g., When mixing socially I am uncomfortable). Items are rated on a 5-point Likert scale from 0 (Not at all) to 4 (Extremely) on how characteristic the statement is to the participant, with higher scores representing higher levels of social anxiety. The SIAS has demonstrated high internal consistency, with alphas greater than .88 in both clinical and non-clinical samples (Mattick & Clarke, 1998; Kählke et al., 2019), as well as good test-retest reliability at 4 and 12 weeks (Mattick & Clarke, 1998). A cut-off score of 34 has reliably differentiated between those with and without a diagnosis of social anxiety disorder (Brown et al., 1997). "In the past week. . ." will be the reference for in the directions for T4 and "In the past month . . . " will be the reference for T5.
Change in PTSD Checklist for DSM-5 (PCL-5; Weathers et al., 2013) | Day 0 (Online baseline survey), Day 7, and one month follow-up (week 5)
  The PCL-5 is a 20-item self-report measure of symptoms of PTSD as defined by the Diagnostic and Statistical Manual, 5th edition (DSM-5). Participants are instructed to keep in mind the worst event they identified on the Life Events Checklist for DSM-5 (LEC-5) when responding to the items. The "past month" version will be used for T1, and T5 and the "past week" version will be used for T4. A total score clinical cut-off of 33 was recommended by Wortmann et al. (2016) for identifying probable PTSD, with 93% sensitivity. The PCL-5 has been identified by the PhenX Toolkit (Hamilton et al., 2011) as a common data element for the assessment and diagnosis of PTSD, and is considered to be well established.
Change in Circumscribed Fear Measure, Most Feared (CFM-MF; McCraw & Valentiner, 2015) | Day 0 (Online baseline survey), Day 7, and one month follow-up (week 5)
  The CFM-MF is a 26-item measure of specific phobia, with subscales that reflect the DSM-5 diagnostic criteria. The measure consists of a screener item (i.e., Please check the box of the object or situation you are most afraid of), which allows for the identification of most feared stimuli, followed by 25 items assessing reactions to the feared stimuli. Participants rate their agreement with each of the 25 statements on 5-point Likert scale from 0 (Strongly disagree) to 5 (Strongly agree), with higher scores reflecting greater fear responding to the most feared stimuli. The CFM-MF has demonstrated high internal consistency (a = .94), as well as good criterion validity with a measure of functional impairment (McCraw & Valentiner, 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Illinois University, DeKalb, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available in the NDA.

REFERENCES:
- [Background] Barrett J, Armony JL. Influence of trait anxiety on brain activity during the acquisition and extinction of aversive conditioning. Psychol Med. 2009 Feb;39(2):255-65. doi: 10.1017/S0033291708003516. Epub 2008 May 9. PMID 18466667
- [Background] Bar-Haim Y. Research review: Attention bias modification (ABM): a novel treatment for anxiety disorders. J Child Psychol Psychiatry. 2010 Aug;51(8):859-70. doi: 10.1111/j.1469-7610.2010.02251.x. Epub 2010 May 6. PMID 20456540
- [Background] Block SR, Liberzon I. Attentional processes in posttraumatic stress disorder and the associated changes in neural functioning. Exp Neurol. 2016 Oct;284(Pt B):153-167. doi: 10.1016/j.expneurol.2016.05.009. Epub 2016 May 10. PMID 27178007
- [Background] Davis M. Neural systems involved in fear and anxiety measured with fear-potentiated startle. Am Psychol. 2006 Nov;61(8):741-756. doi: 10.1037/0003-066X.61.8.741. PMID 17115806
- [Background] Eysenck MW, Derakshan N, Santos R, Calvo MG. Anxiety and cognitive performance: attentional control theory. Emotion. 2007 May;7(2):336-53. doi: 10.1037/1528-3542.7.2.336. PMID 17516812
- [Background] Lazarov A, Suarez-Jimenez B, Abend R, Naim R, Shvil E, Helpman L, Zhu X, Papini S, Duroski A, Rom R, Schneier FR, Pine DS, Bar-Haim Y, Neria Y. Bias-contingent attention bias modification and attention control training in treatment of PTSD: a randomized control trial. Psychol Med. 2019 Oct;49(14):2432-2440. doi: 10.1017/S0033291718003367. Epub 2018 Nov 12. PMID 30415648
- [Background] Pacheco-Unguetti AP, Acosta A, Marques E, Lupianez J. Alterations of the attentional networks in patients with anxiety disorders. J Anxiety Disord. 2011 Oct;25(7):888-95. doi: 10.1016/j.janxdis.2011.04.010. PMID 21641180
- [Background] Sehlmeyer C, Dannlowski U, Schoning S, Kugel H, Pyka M, Pfleiderer B, Zwitserlood P, Schiffbauer H, Heindel W, Arolt V, Konrad C. Neural correlates of trait anxiety in fear extinction. Psychol Med. 2011 Apr;41(4):789-98. doi: 10.1017/S0033291710001248. Epub 2010 Jun 16. PMID 20550755
- [Background] Taylor CT, Cross K, Amir N. Attentional control moderates the relationship between social anxiety symptoms and attentional disengagement from threatening information. J Behav Ther Exp Psychiatry. 2016 Mar;50:68-76. doi: 10.1016/j.jbtep.2015.05.008. Epub 2015 May 23. PMID 26072705
- [Background] Bush G, Shin LM, Holmes J, Rosen BR, Vogt BA. The Multi-Source Interference Task: validation study with fMRI in individual subjects. Mol Psychiatry. 2003 Jan;8(1):60-70. doi: 10.1038/sj.mp.4001217. PMID 12556909